CLINICAL TRIAL: NCT05920785
Title: Clinical and Metabolic, Immunological and Microbiological Characteristics as the Basis of Differentiated Management Tactics for Obese Children
Brief Title: Clinical and Metabolic, Immunological and Microbiological Characteristics of Obese Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 9832
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Obesity
Keywords: childhood obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Occult Blood; Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Blood serum to determine the level of interleukins
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Metabolically healthy obesity: Patients diagnosed with "exogenous constitutional obesity", but without complications of this disease
  Interventions: Diagnostic Test: Determination of the level of interleukins in the blood, stool analysis for the intestinal microbiome, general clinical tests, glucose tolerance test, hormonal profile
- Metabolically unhealthy obesity: Patients diagnosed with "Exogenous constitutional obesity" with the presence of complications of this disease: arterial hypertension, dyslipidemia, impaired carbohydrate metabolism, type 2 diabetes hyperuricemia
  Interventions: Diagnostic Test: Determination of the level of interleukins in the blood, stool analysis for the intestinal microbiome, general clinical tests, glucose tolerance test, hormonal profile
- Control group: Healthy children with normal body weight
  Interventions: Diagnostic Test: Determination of the level of interleukins in the blood, stool analysis for the intestinal microbiome, general clinical tests, glucose tolerance test, hormonal profile

INTERVENTIONS:
Diagnostic Test: Determination of the level of interleukins in the blood, stool analysis for the intestinal microbiome, general clinical tests, glucose tolerance test, hormonal profile — comprehensive laboratory and instrumental diagnostics in accordance with federal clinical guidelines on obesity (Peterkova V. A., 2021), including:
  * general blood test, general urine test,
  * biochemical blood analysis (total protein, urea, creatinine, total bilirubin, AST, ALT, total cholesterol, high and low density lipoproteins, triglycerides, uric acid, alkaline phosphatase, C-reactive protein),
  * hormonal profile (T4 free, TSH, cortisol, C-peptide, fasting insulin, stimulated insulin),
  * glycated hemoglobin,
  * - glucose tolerance test,
  * ultrasound examination of abdominal organs, kidneys (in the presence of arterial hypertension),
  * blood pressure monitoring.
  Special laboratory methods:
  * Blood test to determine the level of HCRP, pro-inflammatory cytokines (leptin, IL-1b, IL-6, IL-8, tumor necrosis factor-α).
  * analysis of feces for microbiota by MALDI-TOF mass spectrometry,
  * bioimpedance measurement.

SUMMARY:
The purpose of the study:

To develop a differentiated management strategy for obese children based on the analysis of the relationship between their clinical, metabolic, immunological and microbiological status

Research objectives:

1. To give a clinical and metabolic characteristic of a group of obese children (age, gender, degree of obesity, body mass index SDS, the presence of complications of obesity, clinical signs of metabolic syndrome, laboratory markers: AlT, AsT, cholesterol, high and low density lipoproteins, uric acid, insulin, leptin).
2. To study the immunological indicators of inflammation in obese children (the level of highly sensitive CRP, proinflammatory cytokines - IL-1b, IL-6, IL-10, IL-18, TNF-α).
3. To assess the state of the intestinal microbiota in obese children by MALDI-TOF mass spectrometry.
4. To analyze the relationship of clinical-metabolic, immunological and microbiological status in obese children and identify markers associated with metabolic syndrome and the formation of complications.

Materials and methods:

At stage 1, it is planned to conduct a cohort study in a group of school-age children with obesity (n=120) with the study of their clinical, metabolic, immunological and microbiological status. The control group will consist of healthy children of the appropriate age who are not overweight (n= 20).

Stage 2 of the study consists in prospective observation of children of the examined group who do not have complications and clinical manifestations of metabolic syndrome for 6 months against the background of standard therapeutic measures (diet, lifestyle correction, physical activity) and repeated clinical and laboratory examination.

DETAILED DESCRIPTION:
The aim of the study:

To develop differentiated management tactics for obese children based on the analysis of the relationship between their clinical, metabolic, immunological and microbiological status.

Research objectives:

1. To give a clinical and metabolic characteristic of a group of obese children (age, gender, degree of obesity, body mass index SDS, the presence of complications of obesity, clinical signs of metabolic syndrome, laboratory markers: AlT, AsT, cholesterol, high and low density lipoproteins, uric acid, insulin, leptin).
2. To study the immunological indicators of inflammation in obese children (the level of highly sensitive CRP, proinflammatory cytokines - IL-1b, IL-6, IL-10, IL-18, TNF-α).
3. To assess the state of the intestinal microbiota in obese children by MALDI-TOF mass spectrometry.
4. To analyze the relationship of clinical-metabolic, immunological and microbiological status in obese children and identify markers associated with metabolic syndrome and the formation of complications.
5. To evaluate the effectiveness of the standard approach to the management of obese children, depending on the characteristics of their clinical, metabolic, immunological and microbiological status, to propose clinical and laboratory predictors of its inefficiency and differentiated management tactics.

The novelty of the study:

For the first time, a comprehensive assessment of the clinical, metabolic, immunological and microbiological status of obese children in the Russian Federation will be carried out. For the first time, the relationship between the level of inflammatory markers, metabolic profile data and the state of the intestinal microbiota, depending on the clinical characteristics of obese patients, will be studied. For the first time, the effectiveness of the standard approach to the treatment of obesity will be analyzed depending on the characteristics of the clinical, metabolic, immunological and microbiological status in obese children.

Practical significance:

Based on the results of the study, metabolic, immunological and microbiological markers associated with the development of complications of childhood obesity and predictors of the ineffectiveness of the standard approach to the management of obese children will be developed, as well as tactics for their differentiated management will be proposed.

Materials and methods:

At stage 1, it is planned to conduct a cohort study in a group of school-age children with obesity (n=120) with the study of their clinical, metabolic, immunological and microbiological status. The control group will consist of healthy children of the appropriate age who are not overweight (n= 20).

Stage 2 of the study consists in prospective observation of children of the examined group who do not have complications and clinical manifestations of metabolic syndrome for 6 months against the background of standard therapeutic measures (diet, lifestyle correction, physical activity) and repeated clinical and laboratory examination.

Inclusion criteria:

1. The presence of a diagnosis of "obesity of egzogenic-constitutional genesis" (according to the criteria of WHO anthropometric standards with the calculation of the standard sigma deviation - SDS using the WHO-AnthroPlus program).
2. The age of children from 7 to 16 years inclusive.
3. Absence of clinically significant concomitant somatic diseases that have a potential impact on the growth, weight and physical development of the child, as well as syndromic or monogenic forms of obesity (Prader-Willi syndrome, Alstrom, etc.)
4. Availability of voluntary informed consent of the legal representative or the child (over 14 years old) for the processing, storage and analysis of personal data the data obtained during the study.

Exclusion criteria:

1. The presence in the anamnesis of any acute infectious diseases, exacerbations of chronic infectious diseases, as well as concomitant diseases affecting the physical development of the child.
2. The presence of syndromic and monogenic forms of obesity.
3. Taking medications that affect the child's appetite (glucocorticosteroids, neuroleptics, antidepressants, etc.).
4. Lack of signed informed consent for inclusion in the study.

Description of the study:

The study includes 2 stages. The first stage includes a general clinical examination of the patient, which includes:

* collection of complaints and anamnesis (life history, family history, endocrinological history),
* features and nature of family and child nutrition,
* assessment of motor activity,
* assessment of the emotional state of the parents and the child,
* general examination data (assessment of the condition of the skin, the type of distribution of subcutaneous fat, the state of the musculoskeletal system, assessment of the stage of puberty, etc.)
* anthropometric parameters (measurement of height and weight, calculation of SDS body mass index, determination of waist/hip ratio index)
* evaluation of the obtained anthropometric data using percentile tables and the WHO-AnthroPlus computer program.

In addition, comprehensive laboratory and instrumental diagnostics will be carried out in accordance with the federal clinical guidelines on obesity (Peterkova V. A., 2021), including:

* general blood test, general urine test,
* biochemical blood analysis (total protein, urea, creatinine, total bilirubin, AST, ALT, total cholesterol, high and low density lipoproteins, triglycerides, uric acid, alkaline phosphatase, C-reactive protein),
* hormonal profile (T4 free, TSH, cortisol, C-peptide, fasting insulin, stimulated insulin),
* glycated hemoglobin,
* glucose-tolerant test,
* ultrasound examination of abdominal organs, kidneys (in the presence of hypertension),
* blood pressure monitoring.

Special laboratory methods:

* a blood test to determine the level of HCRP, pro-inflammatory cytokines (leptin, IL-1b, IL-6, IL-8, tumor necrosis factor-α).
* analysis of feces for microbiota by MALDI-TOF mass spectrometry,
* bioimpedance measurement. The results of the examination will be processed to identify the relationship of the clinical, metabolic, immunological and microbiological status of obese children with their clinical characteristics (degree of obesity, age, sex of SDS body mass index, complications of obesity).

Statistical processing of the received data will be carried out using the Statistica software package. The systematization of the data will be given in the form of a standard deviation (M ±SD). The statistical significance of the differences will be made using the calculated Mann-Whitney U-test. The relationship between the studied features and parameters will be evaluated using Pearson chi-square. The differences will be considered statistically significant at p<0.05.

Depending on the results of the examination, patients will be given recommendations on lifestyle changes and the nature of nutrition aimed at reducing body weight, according to federal clinical guidelines.

Before the second stage of the study, children who do not require pathogenetic therapy to correct complications of obesity (i.e., who do not have impaired carbohydrate metabolism, severe insulin resistance or type 2 diabetes mellitus) will be admitted. The second stage of the study will include two visits - 3 and 6 months after discharge from the hospital, during which the following:

* general examination (assessment of the condition of the skin, the type of distribution of subcutaneous fat, assessment of the stage of puberty, etc.),
* assessment of the emotional state of the child,
* measurement of anthropometric parameters (measurement of height and weight, calculation of BMI, measurement of waist and hip circumference),
* evaluation of the obtained anthropometric data using percentile tables and the WHO-AnthroPlus computer program,
* analysis of the blood pressure monitoring diary,
* assessment of patient compliance,
* correction of recommendations for lifestyle changes, the nature of nutrition, if necessary, correction of drug therapy.

All patients, regardless of the achieved result in weight loss, will also undergo a repeated laboratory examination, the volume of which corresponds to the volume of studies at stage 1.

All received data will also be subjected to statistical processing.

Research hypothesis:

Identification of a positive correlation of individual indicators of clinical and metabolic (visceral fat level, percentage of fat according to bioimpedance, cholesterol, low and high density lipoproteins, AlT, AsT, uric acid), immunological (HCRP, leptin, IL-1b, IL-6, IL-10, IL-18, TNF-α) and microbiological status (or their associations) with weight, SDS body mass index, the presence of complications of obesity, as well as the ineffectiveness of the standard approach to the management of children during the observation process.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of a diagnosis of "obesity of egzogenic-constitutional genesis" (according to the criteria of WHO anthropometric standards with the calculation of the standard sigma deviation - SDS using the WHO-AnthroPlus program).
2. The age of children from 7 to 16 years inclusive.
3. Absence of clinically significant concomitant somatic diseases that have a potential impact on the growth, weight and physical development of the child, as well as syndromic or monogenic forms of obesity (Prader-Willi syndrome, Alstrom, etc.)
4. The availability of voluntary informed consent of the legal representative or a child (over 14 years old) for the processing, storage and analysis of personal data obtained during the study.

Exclusion Criteria:

1. The presence in the anamnesis of any acute infectious diseases, exacerbations of chronic infectious diseases, as well as concomitant diseases affecting the physical development of the child.
2. The presence of syndromic and monogenic forms of obesity.
3. Taking medications that affect the child's appetite (glucocorticosteroids, neuroleptics, antidepressants, etc.).
4. Lack of signed informed consent for inclusion in the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: a group of obese school-age children (n=120) with the study of their clinical, metabolic, immunological and microbiological status. The control group will consist of healthy children of the appropriate age who are not overweight (n= 20).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
increased levels of interleukins | 02.04.2024 - 15.12.2024
  in patients with metabolic unhealthy obesity, there is an increase in inflammatory markers in the blood serum

CONTACTS AND LOCATIONS:
Overall Officials: Natalia B Migacheva, PhD, Study Director — Samara State Medical University
Locations (1):
- Samara State Medical University, Samara, Samara Oblast, Russia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT05920785/Prot_000.pdf